CLINICAL TRIAL: NCT06109441
Title: Phase 2a, Multicenter, Open-Label Study Evaluating the Efficacy and Safety of ALTB-268 in Subjects With Moderately to Severely Active Ulcerative Colitis Refractory to Biologic Therapy
Brief Title: Efficacy/Safety of ALTB-268 in Subjects w/Moderately to Severely Active UC Refractory to Biologics
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AltruBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTB-268-201
Record Dates: First submitted 2023-10-06; First posted 2023-10-31 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Efficacy; Safety
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALTB-268 (Other): ALTB-268 IP will be administered via subcutaneous injection. One loading dose will be followed by 10 weekly doses of ALTB-268 in the 12 weeks induction study phase. Additional 20 biweekly doses of ALTB-268 will be administered in the 40 week maintenance study period.
  Interventions: Biological: ALTB-268

INTERVENTIONS:
Biological: ALTB-268 — ALTB-268 drug product (DP) for SC injection is supplied as a sterile and preservative-free frozen solution or lyophilized powder. All excipients used in the DP formulation are of multi-compendial quality and have precedence for use in parenteral products.

SUMMARY:
ALTB-268-201 is a Phase 2a, multicenter, single arm, multiple-dose, open-label study evaluating the efficacy and safety of ALTB-268 in subjects with moderately to severely active UC. The study consists of a Screening Phase, an Induction Phase, a Maintenance Phase, and an OLE.

DETAILED DESCRIPTION:
ALTB-268-201 is a Phase 2a, multicenter, single arm, multiple-dose, open-label study evaluating the efficacy and safety of ALTB-268 in subjects with moderately to severely active UC.

The study consists of a Screening Phase, an Induction Phase, a Maintenance Phase, and an OLE. Upon successful completion of the Screening Phase, subjects will return to the clinic for their first visit, which must occur within 28 days of the initial Screening Visit. Eligible subjects will be enrolled to receive a SC loading dose of ALTB-268, followed by a weekly maintenance dose of ALTB-268 in the 12-week Induction Study Phase. Participants entering the maintenance study phase will continue to receive the SC dose of ALTB-268 every two weeks, up to week 52. Upon completion of the maintenance study phase, study participants will be asked to return for an end of study visit in approximately 4 weeks unless they continue in an open-label extension (OLE).

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants 18 to 75 years old, inclusive, at Screening.
2. Willing to provide informed consent and to be compliant with the schedule of study visits and protocol assessments.
3. Diagnosis of UC established at least 12 weeks prior to Screening by standard clinical and endoscopic evidence and corroborated by a histopathology report.
4. Moderately to severely active UC, at the time of Screening, defined as a modified Mayo Score (mMS) of 5-9, inclusive, with an endoscopic subscore of ≥ 2 (from central reading), and a rectal bleeding (RB) subscore of ≥ 1.
5. Evidence of active UC, extending proximal to the rectum with ≥ 15 cm of involved colon.
6. Stable doses of concomitant medications:

   1. Subjects receiving oral corticosteroids for the treatment of UC must be on a stable dose of ≤ 20 mg/day (prednisone or equivalent), or ≤ 9 mg/day budesonide. This dose must be stable from the initial Screening visit until the end of the Induction Phase.
   2. Subjects receiving oral 5-aminosalicylic acid (5-ASA) must be on a stable dose from the initial Screening visit until the end of study.
   3. Subjects receiving immunosuppressants (azathioprine, 6-mercaptopurine [6-MP] or methotrexate) must be on a stable dose for 4 weeks prior to Screening until the end of study treatment. Subjects taking methotrexate are also advised to take folic acid 5 mg/week (or equivalent) if there is no contraindication.
   4. Subjects receiving probiotics must be on a stable dose from the initial Screening visit until the end of study.
   5. Subjects receiving an anti-diarrhetic must be on a stable dose for ≥ 2 weeks prior to Screening until the end of study.
7. Previous treatment with one or two advanced therapy that demonstrated an inadequate response and/or loss of response.
8. Negative pregnancy test during Screening and Day 1 (V0) in females of childbearing potential.
9. Females with reproductive potential must be sexually abstinent or be willing to use a highly effective method of contraception from study start to ≥ 3 months after the final dose of the study drug. Highly effective methods of contraception include:

   1. Hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants); male partner should use a condom;
   2. Intrauterine device or system; or
   3. Surgical sterilization or partner sterile (must have documented proof).
10. Male subjects must be either surgically sterile (must have documented proof), agree to be sexually abstinent, or use a double-barrier method of birth control (e.g., condom and diaphragm with spermicide, condom with cervical cap and spermicide) from first study drug administration to ≥ 3 months after the final dose administration.
11. Male subjects must agree to refrain from donating sperm from first study drug administration to ≥ 3 months after final dose administration.

Exclusion Criteria:

1. Diagnosis of Crohn's colitis, colitis yet to be classified, ischemic colitis, nonsteroidal anti-inflammatory drug (NSAID)-induced colitis, idiopathic colitis (i.e., colitis not consistent with UC), or radiation-induced colitis.
2. Ulcerative colitis limited to the rectum (ulcerative proctitis).
3. Presence of short bowel syndrome.
4. History of colectomy, or presence of an ileostomy or colostomy.
5. History of, or active colonic mucosal dysplasia.
6. Treatment with any intravenous (IV) corticosteroid or rectal therapy during the Screening period.
7. Treatment with any calcineurin inhibitor (e.g., cyclosporine, tacrolimus) from the initial Screening visit.
8. Treatment with NSAIDs within 4 weeks prior to Screening. Short-term use (<7 days) of NSAIDs for non-UC related symptoms is allowed.
9. Treatment with tofacitinib or other Janus Kinase (JAK) inhibitors from the initial Screening visit.
10. Treatment with sphingosine-1-phosphate receptor (S1PR) modulators from the initial Screening visit.
11. Biologic therapy within 56 days or 5 half-lives (whichever is longer) prior to Screening. Confirmation of undetectable or non-therapeutic serum levels, as assessed by the Investigator, will allow for eligibility.
12. Tube feeding, defined formula diets, or parenteral alimentation/nutrition within 3 weeks of first dosing.
13. Treatment with oral antibiotics within 4 weeks prior to Screening or IV antibiotics within 8 weeks prior to Screening.
14. Vaccination with a live or live-attenuated vaccine within 4 weeks prior to Screening.
15. History of dysplasia or malignancy in the past 5 years, except completely excised basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
16. Subjects with a current or recent history of severe, progressive, or uncontrolled cardiac (including uncontrolled hypertension), renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, or neurological (e.g., history of seizures) disease, or any other severe comorbidity that, in the opinion of the Investigator, could confound the study results or put the subject at unreasonable risk.
17. Significant screening electrocardiogram (ECG) abnormalities, including evidence of acute myocardial infarction, complete left bundle branch block, second-degree heart block, or complete heart block.
18. For males, a QTc interval (Fridericia's correction) of >450 ms, and for females, a QTc interval (Fridericia's correction) of >470 ms.
19. Any of following laboratory abnormalities during the Screening period. If values are initially outside prescribed limits, the evaluation may be repeated once within the Screening period to determine eligibility:

    1. Calculated creatinine clearance < 60 mL/min
    2. Serum transaminases > 2.0x Upper Limit Normal (ULN)
    3. Alkaline phosphatase (ALP) > 2.0x ULN
    4. Bilirubin > 1.5x ULN; does not apply to subjects with Gilbert's Syndrome (Meulengracht Syndrome)
    5. Hemoglobin < 8g/dL
    6. Platelets < 75,000/μL
    7. Absolute neutrophil count < 1,500/ μL
    8. Absolute lymphocyte count < 800/ μL
20. Human immune deficiency virus (HIV) infection or known HIV-related malignancy.
21. Acute or chronic hepatitis B (HBV) or hepatitis C (HCV), or carrier status. Subjects with anti-HBc (hepatitis B core) antibodies (Ab) but with undetectable anti-HBs (hepatitis B surface) Ab should be excluded.
22. Positive immunoglobulin M (IgM) Ab titers in the presence of negative immunoglobulin G (IgG) Ab titers to Epstein-Barr virus (EBV).
23. Positive stool test for ova or parasites, positive stool culture for pathogens, or positive stool toxin assay for Clostridium difficile at Screening.
24. Active cytomegalovirus (CMV) infection at Screening, as assessed by the Investigator.
25. Positive QuantiFERON® TB test at Screening for latent Mycobacterium tuberculosis (TB) infection. If a QuantiFERON® TB test is indeterminate, the test should be repeated. If the result is again indeterminate, the subject should be excluded.

    Subjects with a history of latent TB infection who received or are receiving an appropriate and documented course of therapy can be included if the screening examination and a chest x-ray performed within 3 months prior to Screening revealed no evidence of current active infection.
26. History of any opportunistic infection within 12 weeks of first dosing.
27. Any current or recent symptoms/signs of infection, except nasopharyngitis, within 4 weeks of first dosing.
28. Cirrhosis or active alcohol abuse, pr the judgment of the Investigator.
29. History of drug abuse according teo the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria within 12 months prior to Screening or a positive drug screening test.
30. Currently breast feeding, or pregnant.
31. Known hypersensitivity or intolerance to ALTB-268 or any of its excipients.
32. Participation in another clinical trial AND having received investigational medication within 30 days or 5 half-lives (whichever is longer) prior to Screening or having used an investigational device treatment within 30 days prior to Screening. Concurrent participation in an observational or long-term follow-up study and not actively receiving an investigational drug or device treatment may be eligible for participation in this study.
33. Inability to comply with the study protocol, in the opinion of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy - change in mMS | week 12
  Change from baseline in mMS at Week 12. The modified Mayo score (mMayo Score) is a measure of disease activity in ulcerative colitis. It is based on stool frequency (SF), rectal bleeding (RB), and endoscopic subscore (ES). The mMS ranges from 0 to 9. A lower mMS means less severe UC, and a higher mMS means more severe UC.

SECONDARY OUTCOMES:
Efficacy - clinical response | week 12 and week 52
  The proportion of subjects with clinical response at Week 12 and Week 52, defined as a decrease from baseline in the mMS of ≥ 2 points AND at least a 30% reduction from the baseline score, AND a decrease in the RB subscore of ≥ 1 point or an absolute RB score of 0 or 1.
Efficacy - clinical remission | week 12 and week 52
  The proportion of subjects with clinical remission at Week 12 and Week 52, defined as mMS of ≤ 2 points, with a SF subscore of ≤ 1 point, a RB subscore of 0, and an endoscopic subscore of ≤ 1 point.
Efficacy - endoscopic improvement | week 12 and week 52
  The proportion of subjects with endoscopic improvement, defined as a centrally read endoscopy score of ≤1 at Week 12 and Week 52.
Efficacy - endoscopic remission | week 12 and week 52
  The proportion of subjects with endoscopic remission, defined as a centrally read endoscopy score of 0 at Week 12 and Week 52
Efficacy - histological remission (RHI) | week 12 and week 52
  Histological remission, defined as a Robarts Histopathology Index (RHI) Score of ≤ 3 at Week 12 and Week 52.
Efficacy- change from baseline in RHI score | week 12 and week 52
  Change from baseline in RHI score at Week 12 and Week 52
Efficacy - Histological remission (Geboes) | week 12 and week 52
  Histological remission, defined as a Geboes score of ≤ 2 at Week 12 and Week 52.
Efficacy - change from baseline in Geboes score | week 12 and week 52
  Change from baseline in Geboes score at week 12 and 52
Efficacy -Change from baseline in mMS | week 52
  Change from baseline in mMS at Week 52
Efficacy - Clinical response and /or clinical remission | week 52
  The proportion of responders who remain in clinical response and/or clinical remission at Week 52.
Efficacy - corticosteroid free clinical remission | week 52
  The proportion of subjects with corticosteroid-free clinical remission at Week 52 in subjects receiving corticosteroids on the first day of dosing and electing to undergo corticosteroid tapering during the Maintenance Phase
Efficacy - corticosteroid free clinical response | week 52
  The proportion of subjects with corticosteroid-free clinical response at Week 52 in subjects receiving corticosteroids on the first day of dosing and electing to undergo corticosteroid tapering during the maintenance phase.
Efficacy - change from baseline in pMS | week 12 and week 52
Efficacy - change in mMS | week 12 and week 52
  Change in individual mMS subscores
Efficacy - change in IBDQ score | week 12 and week 52
  Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) score at Week 12 and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: David Lin, MD, PhD, Study Director — AltruBio Inc.
Locations (24):
- United States (23):
  - San Diego Gastroenterology, San Diego, California
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - Gastro Health Research, Miami, Florida
  - Digestive and Liver Center of Florida, LLC, Orlando, Florida
  - Alliance Clinical Research of Tampa, LLC., Tampa, Florida
  - Gastro Health Partners Southern Indiana, New Albany, Indiana
  - Gastro Health Partners Louisville, Louisville, Kentucky
  - Louisiana Research Center, LLC., Shreveport, Louisiana
  - Gastroenterology Associates of North Mississippi, Oxford, Mississippi
  - New York Presbyterian Hospital - Weill Cornell Medical Colllege, New York, New York
  - Gastroenterology Group of Rochester, Rochester, New York
  - Digestive Disease Medicine of Central New York, Utica, New York
  - Dayton Gastroenterology, LLC, Beavercreek, Ohio
  - Gastro Health Ohio, Liberty Township, Ohio
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Gastroenterology Associates, P.A., Greenville, South Carolina
  - DHAT / GI Aliance, Garland, Texas
  - Caprock Gastro Reasearch, Lubbock, Texas
  - GI Alliance, Mansfield, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - Tyler Research Institute, Tyler, Texas
  - GI Alliance, Webster, Texas
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Wellness Clinical Research, LLC, Vega Baja, Puerto Rico

IPD SHARING:
Plan to Share IPD: No